CLINICAL TRIAL: NCT01302886
Title: A Single-arm, Open-label, Phase 2 Clinical Trial Evaluating Disease Response Following Treatment With Intravenous BHQ880, a Fully Human, Anti-Dickkopf1 (DKK1) Neutralizing Antibody in Previously Untreated Patients With High-risk, Smoldering Multiple Myeloma
Brief Title: Study of BHQ880 in Patients With High Risk Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBHQ880A2204; 2010-022029-13 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-02-24 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-02

CONDITIONS: Smoldering Multiple Myeloma
Keywords: High risk Smoldering multiple myeloma,; BHQ880,; MM
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — BHQ880

ARMS (1):
- BHQ880 (Experimental)
  Interventions: Drug: BHQ880

INTERVENTIONS:
Drug: BHQ880

SUMMARY:
This study will assess the antimyeloma effects of BHQ880A in patients with smoldering multiple myeloma with high risk of progression to active multiple myeloma. BHQ880 will be administered every 28 days in previously untreated patients. Disease assessments will be performed monthly and effects on bone metabolism will be assessed by measurement of serum and urine bone biomarkers, changes in BMD , and QCT with FEA. Additionally, the PK profile of BHQ880 as a single agent and following multiple doses will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of SMM with high-risk for progression to multiple myeloma

   1. BMPC ≥ 10% and serum M-protein level ≥ 3 g/dL, OR
   2. BMPC ≥ 10%, serum M-protein level < 3 g/dL, and an abnormal free light chain ratio of < 0.125 or > 8.0
2. No previous or current anti-myeloma therapies
3. Patients ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 1

Exclusion Criteria:

1. Previous treatment with IV bisphosphonates (i.e., pamidronate or zoledronic acid
2. Another primary malignant disease that requires systemic treatment
3. Concomitant Paget's disease of bone, uncorrected hyperparathyroidism, or uncontrolled thyroid disease
4. Clinically significant uncontrolled heart disease (e.g., unstable angina, congestive heart failure, uncontrolled hypertension, ventricular or atrial arrhythmias)
5. Treatment with an investigational product within 28 days before the first dose of study treatment
6. Pregnant or nursing (lactating) women
7. Women of child-bearing potential, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (Complete Response + Partial Response + Minimal Response) of patients achieving an objective response (defined according to the IMWG uniform response criteria by the Frequency of response of serum or urine M-protein to BHQ880A | at 6 month

SECONDARY OUTCOMES:
Safety and tolerability of BHQ880 in patients with smoldering multiple myeloma by assessing AEs, SAEs, clinical laboratory values | From start of study until disease progression
Characterize the PK profile of BHQ880 as a single agent administered monthly by assessing BHQ880 levels in plasma | Throughout the study until disease progression
Evaluate the effect of BHQ880 on bone metabolism by assessing serum and urine bone biomarkers | Throughout the study until disease progression
Evaluate the effect of BHQ880 on bone mineral density by DXA scan and QCT | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (10):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - H. Lee Moffitt Cancer Center & Research Institute SC - 3, Tampa, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Hematology (2), Atlanta, Georgia
  - Indiana University Indiana Univ, Indianapolis, Indiana
  - Dana Farber Cancer Institute DFCI (2), Boston, Massachusetts
  - Washington University School of Medicine Dept. of WUSTL, St Louis, Missouri
  - Hackensack University Medical Center Multiple Myeloma Division, Hackensack, New Jersey
  - Mount Sinai School of Medicine Mt Sinai, New York, New York
  - Duke University Medical Center Duke SC, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center Fred Hutchinson, Seattle, Washington
- Novartis Investigative Site, Lille, France
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg

REFERENCES:
- See also: Results for CBHQ880A2204 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12765